CLINICAL TRIAL: NCT00005979
Title: Phase III Randomized Study of Intensive Adjuvant Chemotherapy for Resected Colon Cancer at High Risk of Recurrence
Brief Title: Combination Chemotherapy With or Without Irinotecan in Treating Patients With Stage III Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067967; FRE-FNCLCC-ACCORD-2; FFCD-9802; EU-20014
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known if combination chemotherapy is more effective with or without irinotecan in treating colon cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without irinotecan in treating patients who have stage III colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of leucovorin calcium and fluorouracil with or without irinotecan on the 3 year survival rate and overall survival of patients with resected node positive colon cancer at high risk of recurrence.
* Compare toxicities of these regimens in these patients.
* Compare quality of life of these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, disease type (occlusion vs perforation vs N2 only), delay between surgery and chemotherapy (28 days or less vs over 28 days), and age (under 65 vs 65 and over). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV over 22 hours on days 1 and 2.
* Arm II: Patients receive irinotecan IV over 90 minutes on day 1 followed by leucovorin calcium and fluorouracil as in arm I.

Treatment repeats every 14 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed before treatment, after 6 and 12 courses, and then at 1 year.

Patients are followed every 3 months for 2 years, then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 400 patients (200 per arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage III adenocarcinoma of the colon that has been curatively resected within past 42 days
* No metastatic disease
* Node positive

  * No more than 4 nodes affected (Tx, N2, M0) AND/OR
  * N1 or N2 with perforation and/or occlusion
* No prior rectal cancer within 10 cm of anal margin or that was treated with preoperative radiotherapy
* No prior inflammatory disease of the intestine

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin less than 1.25 times upper limit of normal (ULN)
* SGOT and SGPT less than 3 times ULN
* Alkaline phosphatase less than 3 times ULN

Renal:

* Not specified

Cardiovascular:

* No myocardial infarction within past 6 months
* No insufficient cardiac function

Other:

* No other serious medical illness
* No active infection
* No other malignancy except skin cancer or carcinoma in situ of the cervix
* No psychological or social condition that would preclude study
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics
* No prior extensive intestinal resection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-07-22 (Actual); Primary Completion 2005-09-26 (Actual); Study Completion 2007-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ychou, MD, PhD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle; Jean Faivre, Study Chair — Federation Francophone de Cancerologie Digestive
Locations (30):
- France (30):
  - Centre Paul Papin, Angers
  - Clinique St. Etienne, Bayonne
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier de Fleyriat, Bourg-en-Bresse
  - Centre Hospitalier de Bourgoin - Jallieu, Bourgoin
  - Centre Hospitalier General, Brivé
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Faculte de Medecine, Dijon
  - Hopital Du Bocage, Dijon
  - Centre Hospitalier Maie Madeleine, Forbach
  - Centre Leon Berard, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Institut Jean Godinot, Reims
  - St Joseph's Medical Center, Reims
  - Centre Hospitalier Universitaire, Reims
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier de Tarbes, Tarbes
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Valence, Valence
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Centre Hospitalier P. Chubert, Vannes
  - Centre Hospitalier Regionale de Vichy, Vichy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Ychou M, Raoul JL, Douillard JY, Gourgou-Bourgade S, Bugat R, Mineur L, Viret F, Becouarn Y, Bouche O, Gamelin E, Ducreux M, Conroy T, Seitz JF, Bedenne L, Kramar A. A phase III randomised trial of LV5FU2 + irinotecan versus LV5FU2 alone in adjuvant high-risk colon cancer (FNCLCC Accord02/FFCD9802). Ann Oncol. 2009 Apr;20(4):674-80. doi: 10.1093/annonc/mdn680. Epub 2009 Jan 29. PMID 19179549
- [Result] Cote JF, Kirzin S, Kramar A, Mosnier JF, Diebold MD, Soubeyran I, Thirouard AS, Selves J, Laurent-Puig P, Ychou M. UGT1A1 polymorphism can predict hematologic toxicity in patients treated with irinotecan. Clin Cancer Res. 2007 Jun 1;13(11):3269-75. doi: 10.1158/1078-0432.CCR-06-2290. Epub 2007 May 17. PMID 17510208